CLINICAL TRIAL: NCT06221059
Title: A Phase II Clinical Study of Efficacy and Safety of HRS-1780 Tablets and Henagliflozin Proline Tablets in the Treatment of Patients With Chronic Kidney Disease (Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Design)
Brief Title: Efficacy and Safety of HRS-1780 Tablets and Henagliflozin Proline Tablets in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS-1780-201
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRS-1780 dose 1 (Experimental)
  Interventions: Drug: HRS-1780 tablet；Henagliflozin Proline tablet；HRS-1780 tablet placebo ；Henagliflozin Proline tablet placebo
- HRS-1780 dose 2 (Experimental)
  Interventions: Drug: HRS-1780 tablet；Henagliflozin Proline tablet；HRS-1780 tablet placebo ；Henagliflozin Proline tablet placebo
- Henagliflozin Proline (Active Comparator)
  Interventions: Drug: HRS-1780 tablet；Henagliflozin Proline tablet；HRS-1780 tablet placebo ；Henagliflozin Proline tablet placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: HRS-1780 tablet；Henagliflozin Proline tablet；HRS-1780 tablet placebo ；Henagliflozin Proline tablet placebo

INTERVENTIONS:
Drug: HRS-1780 tablet；Henagliflozin Proline tablet；HRS-1780 tablet placebo ；Henagliflozin Proline tablet placebo — Drug：HRS-1780 tablet Drug：Henagliflozin Proline tablet Drug：HRS-1780 tablet placebo Drug：Henagliflozin Proline tablet placebo

SUMMARY:
The objective of this study was to evaluate the efficacy of HRS-1780 tablets or Henagliflozin Proline tablets in patients with chronic kidney disease by evaluating UACR change from baseline to Week 13

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-75 years old
2. Body mass index (BMI) ≥18.0 and <50.0 kg/m2 at the screening visit
3. Subjects treated with an angiotensin-converting enzyme inhibitor (ACEI) and/or angiotensin receptor blocker (ARB) for at least 3 months without any adjustments to this therapy for at least 4 weeks prior to the screening visit
4. Diagnosed with chronic kidney disease, and the estimated glomerular filtration rate (eGFR) was ≥30 and <90 mL/min/1.73 m2 calculated using the CKD-EPI formula at the screening visit
5. Urinary albumin/creatinine ratio (UACR) was ≥300 and <3000 mg/g for at least 2 times on different days detected by the local laboratory; at the screening visit
6. HbA1c <9.0% at the screening visit

Exclusion Criteria:

1. A known or suspected allergy to the investigational drug or its components or excipients;
2. Receive a potent inhibitor/inducer of cytochrome P450 3A4 (CYP3A4) within 7 days prior to screening;
3. Within 4 weeks before screening, the following drugs could not maintain the stable regimen: diabetes drugs, hypertension drugs, non-steroidal anti-inflammatory drugs, endothelin receptor antagonists;
4. Receive SGLT-2 or SGLT-1/2 inhibitors within 4 weeks before screening
5. Received glucagon-like peptide-1 receptor agonist (GLP-1RA) within 8 weeks before screening
6. Received systemic glucocorticoid therapy within 3 months before screening
7. Received immunosuppressive drugs or biological agents
8. Received any other study drug treatment within 3 months or 5 half-lives prior to screening
9. Severe hypertension that was not controlled at screening visit or random visit (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg), or systolic blood pressure <90 mmHg
10. Have urinary tract infection or/and genital infection at the screening visit or random visit, or have a history of repeated urinary tract infection or/and genital infection
11. Diagnosed or suspected polycystic kidney disease, lupus nephritis, anti-neutrophil cytoplasmic antibody (ANCA) -associated vasculitis, acute glomerulonephritis, bilateral renal artery stenosis;
12. Acute kidney injury or dialysis treatment within 6 months before screening
13. Received kidney transplant, or plan to receive kidney transplant during the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2024-03-02 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to Week 13 in UACR | From Baseline to Week 13

SECONDARY OUTCOMES:
Change From Baseline to Week 13 in UACR category （>20%, >30%, >40%) | From Baseline to Week 13
Change From Baseline to Week 4, Week 7 in UACR | From Baseline to Week 4, Week 7
Change From Baseline to Week 13 in 24-hour urinary protein quantification | From Baseline to Week 13
Change From Baseline to Week 13 in estimated glomerular filtration rate (eGFR). An eGFR was calculated based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. | From Baseline to Week 13
Change From Baseline to Week 13 in blood pressure | From Baseline to Week 13

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Eastern Theater Command, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided